CLINICAL TRIAL: NCT07391202
Title: Effectiveness of Non-Surgical Mechanical Therapy of Peri-Implantitis With or Without Prosthetic Crown Removal: A Randomized Controlled Trial
Brief Title: Crown Removal in Non-Surgical Peri-Implantitis Therapy: A Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29012026
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Crowns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical therapy with prosthetic crown removal (Experimental): Implants allocated to this group will receive non-surgical peri-implant therapy after temporary removal of the prosthetic crown. The crown will be unscrewed before treatment to allow direct access and full visibility of the implant surface and peri-implant tissues. Mechanical debridement will then be performed under local anesthesia using sonic and ultrasonic devices with dedicated thin tips and Gracey curettes, according to the EFP S3-level clinical practice guidelines. After completion of debridement and biofilm removal, the prosthetic crown will be reinstalled. Patients will receive oral hygiene instructions and reinforcement.
  Interventions: Procedure: Non-Surgical Peri-Implant Therapy without Crown
- Non-surgical therapy without prosthetic crown removal (Active Comparator): Implants allocated to this group will receive non-surgical peri-implant therapy with the prosthetic crown left in place. Mechanical debridement will be performed under local anesthesia using the same instruments and protocol as in the test group (sonic scaler, ultrasonic devices, and Gracey curettes), but with access limited by the presence of the restoration. Professional oral hygiene instructions and reinforcement will also be provided.
  Interventions: Procedure: Non-Surgical Peri-Implant Therapy with Crown

INTERVENTIONS:
Procedure: Non-Surgical Peri-Implant Therapy without Crown — In this group, the prosthetic crown will be temporarily removed before treatment to allow direct and complete access to the peri-implant tissues and implant surface. After local anesthesia, a thorough mechanical debridement will be performed up to the bottom of the peri-implant pocket using sonic scalers, piezoelectric/ultrasonic devices with dedicated thin tips, and Gracey curettes. The absence of the crown enables improved visualization, more effective instrumentation, and more accurate disruption of the submucosal biofilm. At the end of the procedure, the prosthetic crown will be repositioned. Standardized oral hygiene instructions and motivation will be provided. This intervention aims to maximize cleaning efficacy by eliminating prosthetic-related access limitations.
  Arms: Non-surgical therapy with prosthetic crown removal
Procedure: Non-Surgical Peri-Implant Therapy with Crown — In this group, non-surgical mechanical therapy will be carried out with the prosthetic crown left in place. After local anesthesia, debridement of the peri-implant pocket will be performed using the same instruments and protocol as in the test group, including sonic scalers, ultrasonic devices with thin tips, and Gracey curettes. The presence of the crown limits access to some peri-implant areas and reflects routine clinical practice. Patients will receive standardized oral hygiene instructions and reinforcement. This intervention represents the conventional non-surgical management of peri-implantitis without removal of the restoration
  Arms: Non-surgical therapy without prosthetic crown removal

SUMMARY:
The aim of this single-blind, randomized controlled clinical trial is to evaluate whether removal of the prosthetic crown influences the clinical effectiveness of non-surgical mechanical therapy in implants affected by peri-implantitis.

The study is designed to compare changes in several clinical and radiographic parameters between baseline and follow-up examinations at 3, 6, and 12 months. The primary outcome measure will be the mean peri-implant probing depth (PIPD). Secondary outcomes will include changes in gingival recession (REC), radiographic marginal bone level (MBL), modified bleeding index (mBI), and additional patient-related variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one implant diagnosed with peri-implantitis (Berglundh et al., 2018);
* Patients with a crown on the implant affected by peri-implantitis that is removable;
* Patients who have not received non-surgical peri-implant therapy in the previous 6 months;
* Patients who have not taken systemic antibiotic therapy in the previous 3 months.

Exclusion Criteria:

* Full-Mouth Plaque Score (FMPS) > 30% at the time of non-surgical therapy;
* Pregnant or breastfeeding women;
* Relevant medical history, in the opinion of the examining clinician, that could affect the outcome of non-surgical peri-implant therapy;
* Smoking patients consuming > 10 cigarettes/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Peri-implant probing depth (PIPD) | From enrollment to the end of treatment at 1 year
  Change in mean peri-implant probing depth (PIPD) at the implant level (measured at 6 sites per implant) from baseline to 3, 6, and 12 months after crown removal.

IPD SHARING:
Plan to Share IPD: Undecided